CLINICAL TRIAL: NCT03787056
Title: Predictive Value of Progastrin Titer at Diagnosis and of Progastrin Kinetics During Treatment in Cancer Patients
Acronym: ONCOPRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL18_0369
Record Dates: First submitted 2018-10-26; First posted 2018-12-26 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Cancer; Breast Cancer; Gastric Cancer; Renal Cancer; Prostate Cancer; Melanoma; Lung Cancer; Hepatocellular Cancer; Colorectal Cancer; Head and Neck Cancer; Pancreatic Cancer; Ovarian Cancer; Glioblastoma; Endometrial Cancer; Bladder Cancer; Esophageal Cancer; B-cell Lymphoma
Keywords: dd; TUMOR MARKER; PROGASTRIN
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Stomach Neoplasms; Kidney Neoplasms; Prostatic Neoplasms; Melanoma; Lung Neoplasms; Liver Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Glioblastoma; Endometrial Neoplasms; Urinary Bladder Neoplasms; Esophageal Neoplasms; Lymphoma, B-Cell | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer patients (Other): 420 patients affected by different types of cancer and treated in a curative or a palliative intent. In total 17 cohorts will be open, including: breast cancer, head and neck carcinomas, renal cell carcinoma, prostate carcinoma, lung carcinoma, hepatocellular carcinoma, colorectal carcinoma, thyroid cancer, pancreatic adenocarcinoma, ovarian adenocarcinoma, glioblastoma, endometrial adenocarcinoma, bladder carcinoma, oesophago-gastric carcinoma, B-cell lymphoma, gastric carcinomas. Patients enrolled in curative intent treatment cohorts will never have been previously treated for their cancer. Patients enrolled in non-curative intent treatment cohorts will have never been treated for their metastatic cancers previously, or have developed advanced/metastatic diseases as relapses of localized cancers previously treated with curative intent therapeutic strategies. Other cohort will be open (stability cohorts) : nychtemer cohort and post-operative kinetic cohort.
  Interventions: Other: Blood draws

INTERVENTIONS:
Other: Blood draws — Blood draws are realized at each steps of patient disease management. The volume of each blood drawn is 25 mL for progastrin measurements and 5 mL for the dosage of the other tumor markers. The frequency depend to the cancer and treatment administered :
  * Baseline at diagnosis : Local radical treatment : within 24h before surgery, within 24h after surgery and at the post-surgery follow up visit
  * Chemotherapy treatment : every 3 or 4 weeks
  * Radiotherapy : start day and at the end of radiation ("end of treatment" visit)
  * Palliative systemic treatment (only palliative cohorts) : every 3 to 12 weeks. Follow until the third progression or change of treatment line, or alternatively up to 5 years after inclusion
  * In case of PD or TOX
  * Follow up: at each visit scheduled (every 3 months) for the first 2 years, then every 6 months for 3 years
  * Relapse : withdrawn from the study and last progastrin measurement. Patient could be enrolled in the non-curative intent cohort

SUMMARY:
Progastrin is a pro-hormone that, in physiological conditions, is maturated in gastrin in G cells of the stomach. The role of the gastrin is to stimulate the secretion of gastric acids during digestion. It is also important for the regulation of cell growth of the gastric mucosal.

In a healthy person, progastrin is not detectable in the peripheral blood. However, progastrin is abnormally released in the blood of patients with different cancers (colorectal, gastric, ovarian, breast, cervix uterus, melanoma…) The gene GAST coding for progastrin is a direct target gene of the WNT/ß-catenin oncogenic pathway. The activation of this oncogenic pathway is an early event in cancer development.

Chronic activation of the WNT/ß-catenin oncogenic pathway occurs in almost all human solid tumors and is a central mechanism in cancer biology that induces cellular proliferation, blocking of differentiation leading to primary tumor growth and metastasis formation.

Progastrin measured in the peripheral blood of patients on treatments, could be a new powerful marker for diagnosis and prognosis at different stages.

ELIGIBILITY:
* Histologically and/or cytologically documented (documentation obtained before or after diagnostic surgical procedure when clinical suspicion is strong), cancers for the following cohorts:

  o Breast carcinomas

  o Gastric carcinomas

  o Renal carcinomas

  o Prostate carcinomas

  o Lung carcinomas: NSCLC and SCLC

  o Hepatocellular carcinomas

  o Colorectal carcinomas
  * Head and neck carcinomas
  * Thyroid cancer
  * Pancreatic carcinomas
  * Ovarian adenocarcinomas
  * Glioblastoma
  * Endometrial adenocarcinomas
  * Bladder carcinoma
  * Superficial Oesophago-gastric carcinomas
  * Diffuse Large B-cell Lymphomas
* Patient older than 18 years.
* Patients who gave its written informed consent to participate to the study
* Patients affiliated to a social insurance regime

Specific inclusion criteria for curative treatment strategy cancer patients:

* Indication of a treatment strategy with curative intent (surgery; radiotherapy; chemotherapy; hormonotherapy; targeted agents…)
* Patient naïve of anticancer treatments for the considered cancer
* A prior anti-cancer treatment is allowed if this treatment was performed with curative intent, and if it did not include systemic chemotherapy, and if a complete remission ≥ 6 months was observed in between the end of treatment and relapse. Previous local treatments for superficial lesions are allowed without any time restriction (for example among others, intravesical treatment for superficial bladder cancer lesions).

Specific inclusion criteria for non-curative treatment strategy cancer patients:

* Indication of a treatment strategy with no curative intent (radiotherapy; chemotherapy; hormonotherapy; immunotherapy; targeted agents, non-curative surgery, …)
* Patient naïve of anticancer treatments in non-curative setting (except for metastatic hormone-sensitive prostate cancer, see specific inclusion criteria).

The following tumor type specific inclusion criteria must be met in addition to the inclusion criteria listed above:

Breast carcinomas

• All cohorts:

* Invasive breast ductal carcinoma, or
* Invasive breast lobular carcinoma

  * Curative intent treatment patient cohort:
* Planned to be treated with surgery, with/without neo-adjuvant and/or adjuvant chemotherapy and/or anti-hormone treatment

Gastric carcinomas

* All cohorts:

  o Intestinal-type adenocarcinoma, or

  o Diffuse cell type adenocarcinoma
* Curative intent treatment patient cohort:

  * Planned to be treated with surgery with/without neo-adjuvant treatment, with/without adjuvant treatment

Renal carcinomas • All cohorts:

* Any histology of renal cancer is accepted (non-clear cell renal cancer could be included)
* A pathology proof of renal cell carcinoma is not necessarily provided if patients present typical radiologic characteristics of renal cancer on imaging

  • Curative intent treatment patients cohort:
* Planned to be treated with partial or total nephrectomy

Prostate carcinomas

* Curative intent treatment patients cohort:

  o Localized prostate cancer with high risk features : StageT2b , T2c or T3 and/or Gleason >= 4+3 and/or PSA >= 20 and/or N+

  o Planned to be treated with radical prostatectomy or radiotherapy (potentially associated with androgen deprivation therapy). Brachytherapy and/or focused ultrasounds are not allowed.
* Non-curative intent treatment patients cohort:

  * Patients with metastatic castration resistant prostate cancer (mCRPC) defined by validated criteria of EAU, planned to be treated with doceteaxel or cabazitaxel or second generation hormone (i.e. abiraterone or enzalutamide). Patients have to be naïve of treatment for the castration resistant mCRPC. Patients that previously received docetaxel or a 1st or 2nd generation hormonotherapy for their hormone-sensitive prostate cancer in metastatic setting can be included.

Lung carcinomas treated by immunotherapy :

• Non-curative intent patients cohort:

o NSCLC stage IV according to 8th TNM classification planned to be treated with immunotherapy, with/ without chemotherapy

Lung carcinomas excluding those treated with immunotherapy:

* Curative intent treatment patients cohort:

  o NSCLC histology only

  o Stage I-II according to 8th TNM classification

  o Stage IIIA-B according to 8th TNM classification

  o Planned to be treated with radical treatment (surgery or radiotherapy with/without concurrent chemotherapy), potentially associated with neo-adjuvant or adjuvant treatment
* Non-curative intent patients cohort:

  * NSCLC or SCLC stage IV according to 8th TNM classification planned to be treated with a first line of chemotherapy, with/without associated treatments except immunotherapy (radiotherapy, targeted therapies…). Immunotherapy can be administrated for the subsequent lines of treatment.

Hepatocellular carcinomas A pathology proof of HCC is not necessarily provided if patients present typical radiologic characteristics of hepatocellular carcinoma on imaging

* Absence or chronic hepatic encephalopathy, absence of refractory ascites

  * Curative intent treatment patients cohort:
* Indication of a treatment strategy with curative intent, except liver transplantation: surgical resection, monopolar radiofrequency ablation for HCC (1 to 3 nodules ≤3 cm) or multibipolar radiofrequency if nodule ≤4 cm).

  • Non-curative intent patients cohort:
* Indication of a treatment strategy with no curative intent: transarterial intra-hepatic chemoembolization, targeted therapies (tyrosine kinase inhibitors or monoclonal antibodies) or immune therapy.

Colorectal carcinomas

• Curative intent treatment patients cohort:

o Lieberkühn adenocarcinoma associated with metastases planned to be treated with peri-operative chemotherapy +/- targeted agent and interval surgery

Head and neck carcinomas

* All cohorts

  o Head and neck squamous cell carcinoma from oral cavity, oropharynx, hypopharynx, larynx
* Curative intent treatment patients cohort:

  o Planned to be treated with a radical treatment (surgery and/or radiotherapy potentially associated with concurrent chemotherapy) with/without neo-adjuvant/adjuvant chemotherapy.
* Non-curative intent treatment patients cohort:

  o De novo metastatic or metastatic/loco-regional relapse planned to be treated with chemotherapy and/or immunotherapy

Thyroid cancer • Curative intent patient cohort o Thyroid carcinoma differentiated, poorly differentiated, papillary, vesicular, Hurthle Cell o For which a iodine treatment is indicated (Iodine treatment will be discussed after surgery. In the case the histological result does not confirm a high risk thyroid cancer, patient will be withdrawn from the study. In the same way, if a iodine treatment is not recommended after surgery, patient will be withdrawn from the study. In both cases, patient will be replaced).

Pancreatic carcinomas

• Curative intent patients cohort:

o Pancreas exocrine adenocarcinoma planned to be treated with initial surgery with/without neo-adjuvant chemotherapy and with/without adjuvant chemotherapy or radiotherapy

Ovarian adenocarcinomas • Non/uncertain curative intent patients cohort:

o 1st platinum-sensitive relapse

* High or low grade epithelial adenocarcinomas or carcinosarcoma
* Planned to be treated with chemotherapy and/or PARP inhibitors based treatment, +/- interval debulking surgery

Glioblastoma • Curative intent patients cohort:

o Planned to be treated with surgical resection, followed by adjuvant temozolomide and radiotherapy

Endometrial adenocarcinomas

* Non-curative intent patients cohort:

  o Type 1 (endometrioid or mucinous) or type 2 endometrial (serous, clear cell, undifferentiated carcinoma and carcinosarcoma) cancers

  o Planned to be treated with non-curative systemic treatment for metastatic or advanced disease

Bladder carcinoma

* Transitional cell carcinoma • Curative intent treatment patients:
* Patients with localized muscle invasive bladder cancer (>=PT2)
* Planned to be treated with neo-adjuvant cisplatin based chemotherapy, or immunotherapy or a combination of chemotherapy and immunotherapy

Superficial Oesophago-gastric cancer • Curative intent patients cohort:

o Superficial oesophago-gastric carcinomas (adenocarcinomas or epidermoid carcinomas) of Stage T1 planned to be treated by endoscopic surgery

Diffuse Large B-Cell Lymphoma (DLBCL)

• Curative intent patients cohort:

o Patients planned to be treated with R-CHOP (Rituximab-Cyclophosphamide, Hydroxyadriamycine, Oncovin, Prednisone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2018-12-04 (Actual); Primary Completion 2028-01-04 (Estimated); Study Completion 2028-01-04 (Estimated)

PRIMARY OUTCOMES:
ROC curve AUC regarding diagnostic accuracy of progastrin levels at baseline in cancer patients compared to non-cancer controls | At baseline
  Progastrin concentration in plasma samples will be measured with an ELISA Kit (CancerREAD LAB) provided by ECS Progastrin.

SECONDARY OUTCOMES:
Longitudinal kinetic of progastrin values during treatments, assessed by modeled kinetic parameters of interest | 6 years
  A nonlinear mixed effect model will be used to model the progastrin measurements done during treatments and follow-up of patients.The effect of each event (chemotherapy, surgery…) on the progastrin value and in the inter-individual variability of production and/or elimination rates of progastrin will be analyzed. Progastrin will be measured by ELISA, and the values will be expressed in pM.
  Measures will be done depending on the treatment received. Chemotherapy, every 3 or 4 weeks. Oral treatments: every 3 to 12 weeks. Surgery or radiotherapy: before and after the treatment. Follow up: concomitantly to the visits scheduled for the regular follow up of the patients.
Nycthemeral and weekly and post-operative progastrin variations | every 3 hours within 24 hours for the Nycthemeral cohort, and every week for 2 or 3 weeks for the weekly cohort
  24 patients will be selected, upon their agreement and serum high levels, to enter in nychtemer (12 patients) or weekly (12 patients) cohorts. For the Nychtemer cohort, progastrin will be assayed at d1 at 8:00 am; 11:00 am; 2:00 pm; 5:00 pm; 8:00 pm and at d2 at 8:00 For the weekly cohort, progastrin will be assayed Day 1; Day 8; Day 15 and +/- Day 22; ideally on the same hour times. Progastrin will be measured by ELISA, and the values will be expressed in pM.
Determinants of progastrin serum values: hepatic function | 6 years
  A nonlinear mixed effect model will be used to correlate individual values of progastrin (expressed in pM) with individual characteristic on the patient (hepatic function, as measured by the concentration of AST, ALT and bilirubin).
  Measures will be done Chemotherapy, every 3 or 4 weeks. Oral treatments: every 3 to 12 weeks. Surgery or radiotherapy: before and after the treatment. Follow up: concomitantly to the visits scheduled for the regular follow up of the patients
Determinants of progastrin serum values: renal function | 6 years
  A nonlinear mixed effect model will be used to correlate individual values of progastrin (expressed in pM) with individual characteristic on the patient (renal function, as measured by creatinin concentration and creatinin clearance).
  Measures will be done Chemotherapy, every 3 or 4 weeks. Oral treatments: every 3 to 12 weeks. Surgery or radiotherapy: before and after the treatment. Follow up: concomitantly to the visits scheduled for the regular follow up of the patients
Determinants of progastrin serum values: age | at the inclusion
  A nonlinear mixed effect model will be used to correlate the individual characteristics of the patient (age and gender) with progastrin concentration at the inclusion.
Determinants of progastrin serum values: gender | at the inclusion
  A nonlinear mixed effect model will be used to correlate genders with progastrin concentrations at the inclusion.
Overall survival | 6 years
  The relationships between the progastrin kinetics during and after treatment and overall survival will be analyzed. Analyses will be performed separately on patients with curative intent treatment and on patients with palliative intent treatment.
  Measures wil be done At the end of the study (6 years for patients enrolled in curative intent and 5 years for patients enrolled in non-curative intent) or alternatively at the occurrence of progression or relapse.
recurrence free survival | 6 years
  The relationships between the progastrin kinetics during and after treatment and recurrence free survival will be analyzed. Analyses will be performed separately on patients with curative intent treatment and on patients with palliative intent treatment.
  Measures wil be done At the end of the study (6 years for patients enrolled in curative intent and 5 years for patients enrolled in non-curative intent) or alternatively at the occurrence of progression or relapse.
progression free survival | 6 years
  The relationships between the progastrin kinetics during and after treatment and progression free survival will be analyzed. Analyses will be performed separately on patients with curative intent treatment and on patients with palliative intent treatment.
  Measures wil be done At the end of the study (6 years for patients enrolled in curative intent and 5 years for patients enrolled in non-curative intent) or alternatively at the occurrence of progression or relapse.
The tumor size at cancer diagnosis | At baseline
  The size of the tumor will be correlated to progastrin concentration at the time of cancer diagnosis
Complete surgery | 6 years
  The ability of progastrin kinetics during the neoadjuvant period to predict the outcome of the surgery (complete or not) will be analyzed by a ROC curve. If applicable.
time to recurrence (for patients enrolled in curative intent cohorts). | 6 years
  The ability of the progastrin kinetics to predict recurrence free survival (curative cohorts), will be based on parameters estimated with a PK/PD model able to characterize the early kinetics of progastrin during and after the end of treatment and during follow up.
time to progression (for patients enrolled in non-curative intent cohorts) | 6 years
  The ability of the progastrin kinetics to predict progression-free survival (non-curative cohorts) will be based on parameters estimated with a PK/PD model able to characterize the early kinetics of progastrin during and after the end of treatment and during follow up
time to death (whenever it occurred) | 6 years
  The ability of the progastrin kinetics to predict time to death will be based on parameters estimated with a PK/PD model able to characterize the early kinetics of progastrin during and after the end of treatment and during follow up
Comparison of the initial values and of the kinetics of other serum tumor markers (CA15-3, CA 19-9, CA125, CEA, PSA, AFP) with those of progastrin | at the baseline
  The ROC AUC will be compared between classical markers and the prograstrin. Logistic regression will be used to combine the classical marker(s) and the progastrin in order to estimate the diagnostic value of the marker combination.
  progastrin, CA15-3, CA19-9, CA125, CEA, PSA and AFP concentration will be measured on blood sample taken at the inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit YOU, MD, Principal Investigator — Hospices Civils de Lyon
Locations (17):
- France (17):
  - Service de NEURO-ONCOLOGIE du Groupement Hospitalier EST, Bron
  - Service d'ONCOLOGIE DIGESTIVE et HEPATOLOGIE de l'hôpital de la Croix-Rousse, Lyon
  - Service d'ONCOLOGIE DIGESTIVE et HEPATOLOGIE de l'Hôpital E. Herriot, Lyon
  - Service d'Oto-Rhino-Laryngologie de l'Hôpital de la Croix-Rousse, Lyon
  - Service d'Urologie de l'Hôpital E. Herriot, Lyon
  - Service de Gynécologie de l'hôpital de la Croix-Rousse, Lyon
  - Service de Gynécologie du Groupement Hospitalier Est, Lyon
  - Service de Pneumologie de l'hôpital de la Croix-Rousse, Lyon
  - Service de Pneumologie du Groupement Hospitalier Est, Lyon
  - Service d'Hématologie de l'Hôpital Lyon Sud, Pierre-Bénite
  - Service d'ONCOLOGIE DIGESTIVE et HEPATOLOGIE du Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Service d'Oncologie médicale du Centre hospitalier Lyon Sud, Pierre-Bénite
  - Service d'Urologie de l'hôpital Lyon Sud, Pierre-Bénite
  - Service de Chirurgie de l'hôpital Lyon Sud, Pierre-Bénite
  - Service de Dermatologie de l'hôpital Lyon Sud, Pierre-Bénite
  - Service de Gynécologie de l'hôpital Lyon Sud, Pierre-Bénite
  - Service de Pneumologie de l'Hôpital Lyon Sud, Pierre-Bénite

REFERENCES:
- [Derived] You B, Couraud S, Ceruse P, Badet L, Paparel P, Durand A, Guillet M, Merle P, Lescuyer G, Philip CA, Ducray F, Pioche M, Karlin L, Lifante JC, Glehen O, Bolze PA, Chauvenet M, Langlois-Jacques C, Subtil F, Piecyk M, Carrot A, Joubert D, Prieur A, Vire B, Calattini S, Payen L. Diagnostic value of the wnt target and cancer-associated blood biomarker hPG80: ONCOPRO case-control prospective study. Biomark Res. 2025 Jul 1;13(1):91. doi: 10.1186/s40364-025-00793-z. PMID 40598473